CLINICAL TRIAL: NCT07109167
Title: The Safety and Efficacy of Benmelstobart Injection in Patients With Advanced Biliary Tract Malignant Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-007
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benmelstobart combined with gemcitabine and cisplatin (Experimental): Benmelstobart 1200mg, intravenous infusion on Day 1;Gemcitabine 1000mg/m², intravenous infusion over 30 minutes on Day 1 and Day 8;Cisplatin 25mg/m², intravenous infusion on Day 1 and Day 8.
  Maintenance dose of study medication:
  Benmelstobart 1200mg, intravenous infusion on Day 1;Gemcitabine 1000mg/m², intravenous infusion over 30 minutes on Day 1 and Day 8
  Interventions: Drug: Benmelstobart combined with gemcitabine and cisplatin

INTERVENTIONS:
Drug: Benmelstobart combined with gemcitabine and cisplatin — Benmelstobart 1200mg, intravenous infusion on Day 1;Gemcitabine 1000mg/m², intravenous infusion over 30 minutes on Day 1 and Day 8;Cisplatin 25mg/m², intravenous infusion on Day 1 and Day 8. Maintenance dose of study medication: Benmelstobart 1200mg, intravenous infusion on Day 1;Gemcitabine 1000mg/m², intravenous infusion over 30 minutes on Day 1 and Day 8

SUMMARY:
Evaluate the progression-free survival (PFS) of benmelstobart combined with gemcitabine and cisplatin in first-line patients with advanced cholangiocarcinoma, and the progression-free survival (PFS) of benmelstobart combined with anlotinib in second-line patients with advanced cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria

Age: 18 to 75 years old, inclusive; of either sex. Histopathologically confirmed unresectable and previously untreated gallbladder cancer or intrahepatic/extrahepatic cholangiocarcinoma, with at least one measurable lesion per RECIST v1.1 criteria. Tissue samples must be provided for biomarker analysis, preferably recently obtained tissue. If recent tissue is unavailable, 5-8 archived 5μm-thick paraffin-embedded sections are acceptable.

ECOG performance status: 0 or 1. Life expectancy ≥12 weeks.

Normal major organ function, defined as meeting the following criteria:

1. Hematological tests:

   1. Hemoglobin (HB) ≥90 g/L (without blood transfusion within 14 days prior).
   2. Absolute neutrophil count (ANC) ≥1.5×10⁹/L.
   3. Platelet count (PLT) ≥80×10⁹/L.
2. Biochemical tests:

   1. Albumin (ALB) ≥30 g/L (without albumin transfusion within 14 days prior).
   2. ALT and AST <2.5×upper limit of normal (ULN); if liver metastases are present, ALT and AST ≤5×ULN.
   3. Total bilirubin (TBIL) ≤1.5×ULN.
   4. Plasma creatinine ≤1.5×ULN; or creatinine clearance (CCr) ≥60 ml/min. Subject voluntarily agrees to participate, signs the informed consent form, and is able to comply with scheduled study visits and procedures.

Female subjects of childbearing potential or male subjects with partners of childbearing potential must use effective contraception throughout the treatment period and for 6 months after treatment completion.

Exclusion Criteria Confirmed allergy to any component of Benmelstobart Injection. Uncontrolled hypertension (systolic blood pressure >140 mmHg and diastolic blood pressure >90 mmHg), coronary heart disease of Grade I or higher, arrhythmia of Grade I or higher (including QTc interval prolongation: males >450 ms, females >470 ms), or heart failure of Grade I or higher; patients with positive urine protein.

Patients with definite gastrointestinal bleeding tendency, including: active local ulcerative lesions with fecal occult blood test (++); history of melena or hematemesis within 2 months.

Coagulopathy (INR >1.5, APTT >1.5×ULN) or bleeding tendency. Multiple factors affecting oral drug absorption (e.g., inability to swallow, nausea, vomiting, chronic diarrhea, intestinal obstruction, etc.).

Patients with central nervous system metastases. Pregnant or lactating women. Patients with other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix).

Patients with a history of psychotropic drug abuse who are unable to abstain or with mental disorders.

Patients who participated in other drug clinical trials within 4 weeks. Patients with abnormal thyroid function. Urine protein ≥++ or 24-hour urine protein >1.0 g. Radiotherapy to target lesions within 4 weeks prior to the first dose of study treatment.

Use of immunosuppressive drugs within 4 weeks prior to the first dose of study treatment, excluding nasal, inhaled, or other topical glucocorticoids or physiological doses of systemic glucocorticoids (i.e., ≤10 mg/day prednisone or equivalent dose of other glucocorticoids).

Administration of live attenuated vaccines within 4 weeks prior to the first dose of study treatment or planned during the study period.

Major surgical procedures (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment, or unhealed wounds, ulcers, or fractures.

Active, known, or suspected autoimmune disease or history of such diseases within the past 2 years (patients with vitiligo, psoriasis, alopecia, or Graves' disease that did not require systemic treatment in the past 2 years, hypothyroidism requiring only thyroid hormone replacement therapy, and type 1 diabetes requiring only insulin replacement therapy are eligible).

Uncontrolled concurrent diseases including but not limited to: HIV infection (HIV antibody positive); active or poorly controlled severe infections.

Symptomatic congestive heart failure (New York Heart Association class II-IV) or symptomatic or poorly controlled arrhythmias.

History of interstitial lung disease. Pregnant or lactating female patients. Known history of primary immunodeficiency. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Outcome Measure | 3 years
  Time from randomization to death from any cause
Objective Response Rate | 2 years
  It refers to the proportion of patients (mainly solid tumors) whose tumor has shrunk to a certain extent and remained there for a certain period of time, including Complete Response (CR) and Partial Response (PR)
Quality of life score | 3 years
  Quantitative scoring system for patients' self-subjective self-assessment of current symptom tolerance

CONTACTS AND LOCATIONS:
Overall Officials: yan hai Liu, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical University

IPD SHARING:
Plan to Share IPD: No